CLINICAL TRIAL: NCT01136304
Title: Retrospective and Prospective Validation of a Disease Severity Score System (DS3) for Adults With Type 1 Gaucher Disease (GD1)
Brief Title: Validating a New Severity Score System for Adults With Type 1 Gaucher Disease (GD1)
Status: Completed | Type: Observational
Sponsor: University Research Foundation for Lysosomal Storage Diseases, Inc. (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Neal J Weinreb. MD, Principal Investigator, University Research Foundation for Lysosomal Storage Diseases, Inc.
Other Study IDs: URFLSD-2010-01
Record Dates: First submitted 2010-05-31; First posted 2010-06-03 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Gaucher Disease
Keywords: Gaucher disease; Imiglucerase; Cerezyme; Severity score
MeSH Terms: conditions — Gaucher Disease | interventions — imiglucerase

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Whole blood Buccal smears
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with Type 1 Gaucher disease (GD1): Adults with GD1 who are cared for at one of the participating research sites whether treatment naive or treated in past or currently with imiglucerase enzyme replacement treatment.
  Interventions: Drug: Imiglucerase

INTERVENTIONS:
Drug: Imiglucerase — Imiglucerase intravenous infusions regardless of dose or schedule of administration.
  Other Names: Cerezyme

SUMMARY:
With the participation of an international consortium of investigators, the investigators will evaluate the validity of a new severity score system called DS3 for adult patients with Gaucher disease. The investigators hypothesize that initial DS3 scores will be predictive of both disease progression and patterns of response including imiglucerase dose sensitivity and completeness and maintenance of response and that sequential DS3 scores will accurately portray either clinical progression of disease or improvement in response to treatment. The investigators will also collect DNA specimens that in future research will be used in conjunction with the DS3 scores to evaluate determinants of the clinical course and the response to treatments for Gaucher disease.

DETAILED DESCRIPTION:
GD1 is a prototypical lysosomal storage disorder and the first disorder to have compelling evidence of successful treatment with enzyme replacement therapy. The common clinical manifestations are hematologic cytopenias, hepatomegaly, splenomegaly, and a spectrum of skeletal pathologies. Disease expression is diverse. The rate and extent of disease progression are variable and often independent of the age at which symptoms are first reported1. Despite a long history of treatment efficacy2, there is significant heterogeneity of response among patients with regard to the maximum improvement in hematologic, visceral, bone, and other manifestations and the dynamic speed of response during therapy1-3. There have been few well-designed studies that comprehensively annotate phenotypic variation over time or measure treatment efficacy and dose response. In part, this is attributable to lack of a validated disease severity scoring system for GD1 to standardize the monitoring of progression and treatment response and to define patient cohorts in clinical studies.

DS3 is a method of expressing an integrated assessment of the burden of disease in a given patient. It can be used to monitor patient status, determine endpoints in clinical studies, classify disease phenotypes and compare patients with the same disease. Although frequently referred to as 'disease severity indices,' DS3 instruments may also include measures of disease activity and damage. DS3s utilize a minimal data set to score the patient in a comprehensive manner. They usually are structured as a group of domains (often according to organ system) that are populated with non-redundant items that are valid, reliable, use feasible, standardized methods of assessment, and that are variably weighted based on associated morbidity and mortality. A DS3 for adult GD1 patients was recently developed and subjected to successful preliminary testing for validity, reliability and feasibility4. With respect to changes over time, a minimal clinically important difference was defined. Construct validity has been partially demonstrated. Using 20 patient profiles from the International Collaborative Gaucher Group (ICGG) Gaucher Registry, the instrument was shown to correlate very well with the "gold standard" clinical global impression scale. However, larger scale testing in a population that is representative of the world wide distribution of GD1 phenotypes (including splenectomy patients) is needed and predictive validity has yet to be determined. Moreover, the DS3 has not yet been correlated with disease-specific measures of response such as achievement of therapeutic goals or broadly used biomarkers. Combining retrospective and prospective analysis, this study is designed to address these issues

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Type 1 Gaucher disease regardless of treatment status who are enrolled in the International Collaborative Gaucher Group (ICCG) Gaucher Registry and who are cared for at one of the participating research sites.

Exclusion Criteria:

* Children under the age of 18 years

  * Patients with Type 3 Gaucher disease
  * Patients who have declined to be enrolled in the ICCG Gaucher Registry
  * Patients not cared for at one of the participating research sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consenting adult patients with type 1 Gaucher disease who are cared for at one of the participating research sites and who are enrolled in the International Collaborative Gaucher Group Gaucher Registry
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2010-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in total DS3 severity score from baseline score | Calculated annually and assessed up to 25 years until either death, withdrawal from the study, or end of study
  The DS3 score is calculated annually from either date of first treatment or, in untreated patients, from date of first enrollment in the ICGG Gaucher Registry

CONTACTS AND LOCATIONS:
Overall Officials: Neal J Weinreb, MD, Principal Investigator — University Research Foundation for Lysosomal Storage Diseases, Inc.
Locations (2):
- United States (2):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Northwest Oncology Hematology Associates PA, Coral Springs, Florida

REFERENCES:
- [Background] Weinreb NJ, Cappellini MD, Cox TM, Giannini EH, Grabowski GA, Hwu WL, Mankin H, Martins AM, Sawyer C, vom Dahl S, Yeh MS, Zimran A. A validated disease severity scoring system for adults with type 1 Gaucher disease. Genet Med. 2010 Jan;12(1):44-51. doi: 10.1097/GIM.0b013e3181c39194. PMID 20027115
- [Result] Weinreb NJ, Finegold DN, Feingold E, Zeng Z, Rosenbloom BE, Shankar SP, Amato D. Evaluation of disease burden and response to treatment in adults with type 1 Gaucher disease using a validated disease severity scoring system (DS3). Orphanet J Rare Dis. 2015 May 22;10:64. doi: 10.1186/s13023-015-0280-3. PMID 25994334
- [Derived] Ganz ML, Stern S, Ward A, Nalysnyk L, Selzer M, Hamed A, Weinreb N. A new framework for evaluating the health impacts of treatment for Gaucher disease type 1. Orphanet J Rare Dis. 2017 Feb 20;12(1):38. doi: 10.1186/s13023-017-0592-6. PMID 28219443